CLINICAL TRIAL: NCT02803554
Title: Young Donor Plasma Transfusion and Age-Related Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ambrosia LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AM-PL-101
Record Dates: First submitted 2016-06-11; First posted 2016-06-17 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Young donor plasma (Experimental): An infusion of plasma derived from donors aged 25 years or younger
  Interventions: Other: Plasma

INTERVENTIONS:
Other: Plasma — Blood plasma from donors aged 25 years or younger

SUMMARY:
The purpose of the study is to evaluate the beneficial effects of infusions of plasma from young donors using blood biomarkers.

DETAILED DESCRIPTION:
Each patient will receive an infusion of plasma derived from a young donor (16-25 years of age). A panel of age-associated biomarkers will be measured before and after treatment.

We have drawn biomarkers from clinical measures of aging and physiology, biomarkers of disease advancement, as well as biomarkers of aging from animal and human studies. These will represent a spectrum of physiologic pathways with evidence-based connections to aging. They include the physiologic processes of inflammation, neurogenesis, stem cell proliferation, blood clotting, immune function, and amyloid plaques. Organ function which will be specifically measured includes the liver, bone marrow, kidneys, pancreas, muscles, cardiovasculature, cerebrovasculature, and the thyroid. Specific disease states connected to these biomarkers include anemia, neutropenia, thrombocytopenia, obesity, diabetes, high cholesterol, elevated risk of cancer, atherosclerosis, dementia, and cataracts.

Visit us at www.ambrosiaplasma.com

ELIGIBILITY:
Inclusion Criteria:

* 35 years of age or older

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-06; Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Blood biomarkers (1/3) | Change from before treatment to 1 month after treatment
  WBC, RBC, Hemoglobin, Hematocrit, MCV, MCH, MCHC, RDW, Platelet Count, MPV, Differential, Albumin, Albumin/Globulin Ratio (calculated), Alkaline Phosphatase, ALT, AST, BUN/Creatinine Ratio (calculated), Calcium, Carbon Dioxide, Chloride, Creatinine with GFR Estimated, Globulin (calculated), Glucose, Potassium, Sodium, Total Bilirubin, Total Protein, Urea Nitrogen, Adiponectin, Alpha-1-Antitrypsin, Alpha-2-Macroglobulin, Alpha-Fetoprotein, Apolipoprotein A-I, Apolipoprotein A-II, Apolipoprotein C-I, Apolipoprotein C-III
Blood biomarkers (2/3) | Change from before treatment to 1 month after treatment
  Apolipoprotein H, Apolipoprotein(a), Beta-2-Microglobulin, Brain-Derived Neurotrophic Factor, C-Reactive Protein, CD40 Ligand, Cancer Antigen 125, Cancer Antigen 19-9, Carcinoembryonic Antigen, Complement C3, EN-RAGE, Eotaxin-1, Epithelial-Derived Neutrophil-Activating Protein 78, Erythropoietin, Factor VII, Ferritin, Fibrinogen, Granulocyte Colony-Stimulating Factor, Granulocyte-Macrophage Colony-Stimulating Factor, Growth Hormone, Haptoglobin, Human Chorionic Gonadotropin beta, Immunoglobulin A, Immunoglobulin E, Immunoglobulin M, Insulin, Intercellular Adhesion Molecule 1, Interferon gamma, Interleukin-1 alpha, Interleukin-1 beta, Interleukin-1 receptor antagonist, Interleukin-10, Interleukin-12 Subunit p40, Interleukin-12 Subunit p70, Interleukin-13, Interleukin-15, Interleukin-16, Interleukin-17, Interleukin-2, Interleukin-23, Interleukin-3
Blood biomarkers (3/3) | Change from before treatment to 1 month after treatment
  Interleukin-5, Interleukin-6, Interleukin-7, Interleukin-8, Leptin, Macrophage Inflammatory Protein-1 alpha, Macrophage Inflammatory Protein-1 beta, Macrophage-Derived Chemokine, Matrix Metalloproteinase-2, Matrix Metalloproteinase-3, Matrix Metalloproteinase-9, Monocyte Chemotactic Protein 1, Myeloperoxidase, Myoglobin, Neuron-Specific Enolase, Plasminogen Activator Inhibitor 1, Prostate-Specific Antigen, Free, Pulmonary and Activation-Regulated Chemokine, Serum Amyloid P-Component, Stem Cell Factor, T-Cell-Specific Protein RANTES, Thrombospondin-1, Thyroid-Stimulating Hormone, Thyroxine-Binding Globulin, Tissue Inhibitor of Metalloproteinases 1, Transthyretin, Tumor Necrosis Factor alpha, Tumor Necrosis Factor beta, Tumor necrosis factor receptor 2, Vascular Cell Adhesion Molecule-1, Endothelial Growth Factor, Vitamin D-Binding Protein, von Willebrand Factor

IPD SHARING:
Plan to Share IPD: No